CLINICAL TRIAL: NCT05595538
Title: A Feasibility Study Assessing the Safety of Multiple Doses of Anti-SARS-CoV-2 Plasma in Mechanically Ventilated Intubated Patients With Respiratory Failure Due to Coronavirus Disease (COVID-19)
Brief Title: Use of Multiple Doses of Convalescent Plasma in Mechanically Intubated Patients With COVID-19
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hospital Regional Dr. Rafael Estévez (Other)
Collaborators: Complejo Hospitalario Dr. Arnulfo Arias Madrid (Other); Hospital Santo Tomas (Other); Hospital Punta Pacífica, Pacífica Salud (Unknown); Insituto Conmemorativo Gorgas de Estudios para la Salud (Unknown); Sociedad Panameña de Hematología (Unknown); Institute of Scientific Research and High Technology Services (INDICASAT AIP) (Unknown); University of Panama (Unknown); Sistema Nacional de Investigación de Panamá (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPH-COVID-19
Record Dates: First submitted 2022-10-07; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: Convalescent plasma; critically ill; SARS-CoV-2; COVID-19; neutralizing antibodies
MeSH Terms: conditions — COVID-19; Critical Illness | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intubated COVID-19 patients admitted to the ICU. (Experimental): Participants intubated who consent immediately before intubation to receive more than one dose of COVID-19 convalescent plasma.
  Interventions: Biological: Multiple doses of anti-SARS-CoV-2 Convalescent Plasma

INTERVENTIONS:
Biological: Multiple doses of anti-SARS-CoV-2 Convalescent Plasma — SARS-CoV-2 Convalescent Plasma(1-2 units; ~300-600 mL with the presence of IgG anti-SARS-CoV-2.
  Other Names: COVID-19 Convalescent Plasma

SUMMARY:
This study will assess the feasibility and safety of administering multiple doses of convalescent plasma to Covid-19 positive patients admitted to the Intensive Care Unit (ICU) receiving mechanical ventilation. Donor plasma will be obtained from Covid-19 recovered patients. All plasma used in this protocol will be collected following the guidelines issued by the Food and Drug Administration (FDA) and the Ministry of Health in Panama.

Every patient recruited will receive one or two plasma units infused on days 0, 2, 4, 6, and 8. The primary objective of this study is feasibility. Feasibility will be assessed based on the proportion of subjects who consent and receive at least one dose of convalescent plasma more than once. The investigators will evaluate the safety and feasibility of this study by accounting for any related adverse event.

The secondary study endpoints are overall survival at days 14, 28, and 60 after the first dose of convalescent plasma. Respiratory status and overall clinical status will be reviewed during follow-up until day nine and on days 14, 28, and 60.

DETAILED DESCRIPTION:
From historical and anecdotal data on convalescent plasma, it seems its administration is safe in cases of coronavirus infection. Now, the high mortality of COVID-19, particularly in elderly and vulnerable persons such as critically ill patients, suggests that the benefits of its use in those at high risk for death outweigh the risks. However, for all cases where convalescent plasma administration is considered, a risk-benefit assessment must be conducted to assess individual variables.

This study proposed the follow-up of 30 intubated patients due to COVID-19 who have been admitted to the ICU and have consented to receive five doses of one or two units of convalescent plasma.

Every patient will have a follow-up from the consent day to day 60. The study team will monitor and record: vital signs, daily ventilatory requirements, and assessment of clinical status, including new medical conditions and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Hospitalized with COVID-19 respiratory symptoms and confirmation via COVID-19 SARS-CoV-2 Real Time-polymerase chain reaction(PCR) testing.
3. Subject or proxy (including by phone) is willing and able to provide written or digital informed consent and comply with all protocol requirements.
4. Intubated
5. Consent to storage of specimens for future testing.

Exclusion Criteria:

1. Contraindication to transfusion (severe volume overload, history of anaphylaxis to blood products).
2. Severe multi-organ failure, and hemodynamic instability.
3. Other documented uncontrolled infections.
4. Severe disseminated intravascular coagulopathy (DIC) needing factor replacement, FreshFrozen Plasma, cryoprecipitate.
5. On dialysis.
6. Active intracranial bleeding.
7. Clinically significant myocardial ischemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who received at least one unit more than one day | 8 days
  Transfusion of multiple doses (up to 5 doses) of 300-600 ml of convalescent plasma from COVID-19

SECONDARY OUTCOMES:
Development of plasma transfusion reaction | 8 days
  presence of any sign or symptoms of plasma transfusion reaction (TACO, TRALI, fever, rash)
Overall Survival | 60 days
  overall survival up to day 60
oxygen Support | 60 days
  type of ventilatory support by days 9, 14, 28, and 60. The options for types of oxygen support are: Mechanical Ventilation, Non/invasive ventilation, and no support needed.
Clinical Status | 60 days
  Change in 7-point ordinal clinical deterioration scale pre-transfusion to Days 1, 3, 7, 9, 14, 28 and 60 post-transfusion. The 7-point ordinal scale measured by: 7-death, 6-ICU patient who requires extracorporeal membrane oxygenation (ECMO) or mechanical ventilation; 5-ICU patient, do not requires ECMO or mechanical ventilation; 4 -hospitalization and requires supplemental oxygen; 3- hospitalization without supplemental oxygen; 2- limitation of activities, discharge from hospital 1- no limitation of activities, discharge from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Aguilar, M.D, Principal Investigator — 1. Complejo Hospitalario Metropolitano Arnulfo Arias Madrid, Caja de Seguro Social
Locations (1):
- 1. Complejo Hospitalario Metropolitano Arnulfo Arias Madrid, Caja de Seguro Social, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No